CLINICAL TRIAL: NCT02983058
Title: PET Imaging Study of Amish and Mennonite Patients With CNTNAP2 Mutations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To obtain funding for a larger study
Sponsor: Jeffrey A. Lieberman, MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey A. Lieberman, MD, Director, New York State Psychiatric Institute, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #7107; NCT02572206 (obsolete NCT alias)
Record Dates: First submitted 2016-08-25; First posted 2016-12-06 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/SPECT and MRI scans (Other): PET/SPECT scan will be used to evaluate the utility of mGluR5 binding as a biomarker of the CNTNAP2 mutation and related mTOR kinase pathway dysregulation. 30 minutes structural MRI will be obtained to permit co-registration of PET images.
  Interventions: Radiation: PET/SPECT Scan; Device: MRI Scan

INTERVENTIONS:
Radiation: PET/SPECT Scan — PET scan will be performed on a mCT scanner
  Other Names: PET
Device: MRI Scan — Structural MRI will be obtained to permit co-registration of PET images
  Other Names: MRI

SUMMARY:
The primary goal of the present study is to evaluate the utility of mGluR5 binding as measured by PET as biomarker of the CNTNAP2 mutation and related mTOR kinase pathway dysregulation.

DETAILED DESCRIPTION:
The investigators will focus on mGluR5 PET binding as a surrogate measure for level of activity of the mTOR kinase pathway. This study is being conducted by the New York State Psychiatric Institute (NYSPI) and will take place at Columbia University Medical Center (CUMC) in New York City and at a research office in Strasburg, PA. Subjects (n=20) with the CNTNAP2 mutation with schizophrenia or a related condition will be recruited from the Amish and Mennonite communities and brought to CUMC for detailed investigation. Affected individuals will be compared to Amish and Mennonite control subjects drawn from the same families but not harboring CNTNAP2 mutations (n=20). The primary measure will consist of mGluR PET binding in DLPFC. In addition, secondary analyses will assess binding in other brain regions such as hippocampus and visual cortex. Exploratory measures, as well as relationships between PET mGluR5 binding and clinical symptomatology, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Meets DSM-5 diagnostic criteria for psychotic disorder, including schizophrenia, schizoaffective disorder or psychotic disorder not elsewhere classified
* Genetic confirmation that patient carries CNTNAP2 mutation
* Of Amish and/or Mennonite descent
* Has a relative willing to be part of the study and this relative will travel with the participant to CUMC in NYC and back to Lancaster, PA
* Stable enough to travel and participate in the study

Control subjects:

* Genetic confirmation that subject does not carry CNTNAP2 mutation
* First-degree or second-degree relative of subject of Amish/Mennonite descent with CNTNAP2 mutation

Exclusion Criteria (for patients and controls):

* Positive urine toxicology for drugs of abuse
* Positive history of severe neurological illness or history of brain trauma
* Positive history of severe medical illness that would increase risk due to PET scan procedure, or interfere with interpretation of research findings
* Low hemoglobin (Hb < 11 g/dL in males, Hb < 10 g/dL in females)
* Lifetime exposure to radiation in the workplace, or lifetime history of participation in nuclear medicine procedures, including research protocols.
* Blood donation within 8 weeks of study
* Presence of clinically significant brain abnormalities
* Female subjects of child-bearing age who are not surgically sterilized and between menarche and 1 year postmenopausal must test negative for pregnancy at the time of enrollment and prior to the PET scan based on a serum pregnancy test. Women who are breast-feeding are also excluded.
* Metal implants, pacemakers, other metal (e.g., shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with the MR scan
* Medicinal patch, unless removed prior to the MR scan
* Patients: current treatment with clozapine and/or medications other than antipsychotics PRN anxiolytics
* Use of the medications that would interfere with mGluR5 binding, including lamotrigine, gabapentin, topiramate, phenobarbital, pregabalin, zonisamide, N-acetylcysteine, D-cycloserine
* Control subjects: lifetime history of antipsychotic or antidepressant use

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sander Markx, MD, Principal Investigator — New York State Psychiatric Institute

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were exclusively recruited from the Amish and Mennonite community in Lancaster, Pennsylvania (PA). All subjects with psychotic spectrum disorder were receiving clinical care at the Clinic for Special Children in Strasburg, PA and identified an unaffected 1st or 2nd degree relative (unaffected subject).
Pre-assignment Details: All subjects (affected and unaffected) who met inclusion/exclusion criteria were included in the study.
Groups:
- Subjects With Psychotic Spectrum Disorders; Unaffected 1st or 2nd Degree Relatives: PET/SPECT scan will be used to evaluate the utility of mGluR5 binding as a biomarker of the CNTNAP2 mutation and related mTOR kinase pathway dysregulation. 30 minutes structural MRI will be obtained to permit co-registration of PET images.
  PET/SPECT Scan: PET scan will be performed on a mCT scanner
  MRI Scan: Structural MRI will be obtained to permit co-registration of PET images
Period: Overall Study
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected 1st or 2nd Degree Relatives
Started | 7 | 5
Completed | 2 | 2
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Baseline population numbers include all participants who signed consent and underwent screening procedures
Groups:
- Subjects With Psychotic Spectrum Disorders: Subjects who met DSM-5 diagnostic criteria for psychotic disorder and had genetic confirmation of carrying CNTNAP2 mutation
- Unaffected Relatives: Unaffected 1st or 2nd degree relatives of subjects who have psychotic spectrum disorder and carries the CNTNAP2 mutation. Unaffected relatives do not carry CNTNAP2 mutation
- Total: Total of all reporting groups
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected Relatives | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Level of mGluR5 PET Binding in Dorsolateral Prefrontal Cortex (DLPFC) in CNTNAP2 Mutation Carriers vs. Comparison Subjects
Description: Outcome measure is total distribution volume (VT) where distribution volume of the non displaceable compartment (VND) plus binding potential (BPP) with respect to the arterial plasma concentration of tracer. VT=VND + BPP
Time Frame: 90 minutes and the comparison will be binding in the specific regions listed (e.g., DLPFC) controlled by binding in the cerebellum/input function
Population: N was not reached and data was not analyzed
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected 1st or 2nd Degree Relatives
Number analyzed (Participants) | 2 | 2
mL/cm^3 | 13.58 (1.27) | 11.12 (0.24)

2. Secondary Outcome: Level of mGluR5 PET Binding in Hippocampus
Description: Evaluate PET mGluR5 binding in other regions of potential relevance, including hippocampus in order to determine ideal regions of interest for future intervention studies by using VT=VND + BPP. VND is assumed to be equal across brain regions and therefore VT will vary across brain regions with mGluR5 concentration.
Time Frame: 90 minutes and the comparison will be binding in the specific regions listed controlled by binding in the cerebellum/input function
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected 1st or 2nd Degree Relatives
Number analyzed (Participants) | 2 | 2
mL/cm^3 | 10.61 (1.60) | 11.29 (0.53)

3. Secondary Outcome: Level of mGluR5 PET Binding in Primary Visual Cortex (Occipital Pole)
Description: Evaluate PET mGluR5 binding in other regions of potential relevance, including primary visual cortex in order to determine ideal regions of interest for future intervention studies as measured by total distribution volume (VT).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected 1st or 2nd Degree Relatives
Number analyzed (Participants) | 2 | 2
mL/cm^3 | 10.50 (0.87) | 8.74 (1.21)

ADVERSE EVENTS:
Time Frame: From time of consent to 30 days after scans
Arm/Group | Subjects With Psychotic Spectrum Disorders | Unaffected 1st or 2nd Degree Relatives
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02983058/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT02983058/SAP_001.pdf